CLINICAL TRIAL: NCT03513289
Title: Collaborative Assessment of ICU Recovery Needs
Acronym: CAIRN
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Principal Investigator, Carla Sevin, Assistant Professor of Medicine, Director of the ICU Recovery Center at Vanderbilt, Vanderbilt University Medical Center
Other Study IDs: 172158
Record Dates: First submitted 2018-03-05; First posted 2018-05-01 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Post-Intensive Care Syndrome
Keywords: ICU delirium; post-intensive care syndrome; critical illness myopathy
MeSH Terms: conditions — postintensive care syndrome | interventions — Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient, Carer, and Clinician Interviews: This group/cohort consists of patients who experienced critical illness and were hospitalized in an ICU setting.
  Interventions: Other: Patient, Carer, and Clinician Interviews

INTERVENTIONS:
Other: Patient, Carer, and Clinician Interviews — Post-ICU follow-up interviews conducted over the phone, lasting between 30-60 minutes.

SUMMARY:
The primary purpose of this study is to better understand the impact of the Society of Critical Care Medicine (SCCM) THRIVE Collaboratives on patients, their families and clinicians.

The investigators have formed an international and interprofessional evaluative team with experts in the field in an effort to explore interactions between survivors and THRIVE. This approach is reflective of the international ethos of SCCM and its collaboratives, with the potential to improve the generalizability of this survivorship research to different health systems.

DETAILED DESCRIPTION:
The aims of this qualitative study are:

1. To identify elements that helped survivors in their recovery, as well as potential obstacles
2. To capture elements of survivorshop that are generalizable, regardless of participation in the THRIVE collaboratives
3. To gain knowledge to be incorporated back into the collaboratives

Patients, family members, and clinicians will be interviewed and their responses analyzed for themes of ICU recovery including elements that patients and families find helpful to recovery, barriers and facilitators to different models of post-ICU support, including peer support and post-ICU clinics, and drivers of improvement in post-ICU care. Patients, carers, and clinicians with a wide variety of survivorship experiences are encouraged to participate, including those who have participated in a THRIVE collaborative support site (peer support or clinic).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who survived a critical illness, and their carers, who were identified by collaborative members or self-identify as having been through a THRIVE Program.
2. Patients who survived a critical illness, and their carers, who did not participate in a THRIVE program.
3. Clinicians directly involved in the care of ICU survivors in the outpatient setting, who have participated in a THRIVE initiative through the Society of Critical Care Medicine.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and caregivers who were identified by collaborative members, or self-identify, as having been through a THRIVE Program, patients and caregivers who did not participate in a THRIVE program, and clinicians directly involved in the care of ICU survivors in the outpatient setting who have participated in a THRIVE initiative through the Society of Critical Care Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Survivorship Experiences from Patients | 18 months
  30-minute audio-taped, semi-structured interviews with patients informing on post-ICU care coordination

SECONDARY OUTCOMES:
Survivorship Experiences from Caregivers | 18 months
  30-minute audio-taped, semi-structured interviews with caregivers informing on post-ICU care coordination
Survivorship Experiences from Clinicians | 18 months
  30-minute audio-taped, semi-structured interviews with clinicians informing on post-ICU care coordination

CONTACTS AND LOCATIONS:
Overall Officials: Carla M Sevin, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States
- Australian and New Zealand Intensive Care Research Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided